CLINICAL TRIAL: NCT03352934
Title: A Phase II, Open-label, Multicenter Trial to Investigate the Clinical Activity and Safety of Avelumab in Patients With Advanced, Metastatic High Grade Neuroendocrine Carcinomas NEC G3 (WHO 2010) Progressive After Chemotherapy
Brief Title: Avelumab Treatment in Patients With Neuroendocrine Carcinomas (NEC G3) Progressive After Chemotherapy
Acronym: AveNEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Matthias M. Weber, Principal Investigator, Johannes Gutenberg University Mainz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-007; 2016-004373-40 (EudraCT Number)
Record Dates: First submitted 2017-11-03; First posted 2017-11-24 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Cancer
Keywords: avelumab; anti-PD-L1; neuroendocrine tumor; NET G3; neuroendocrine carcinoma; NEC G3
MeSH Terms: conditions — Neoplasms; Neuroendocrine Tumors; Carcinoma, Neuroendocrine | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avelumab (Experimental): 10 mg/kg Avelumab every 2 weeks
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Avelumab will be administered as intravenous infusion at 10 mg/kg once every two weeks until documented disease progression (PD), unacceptable toxicity, or any criterion for treatment withdrawal are met.
  Other Names: MSB0010718C; anti-PD-L1

SUMMARY:
The purpose of the AveNEC trial is to investigate the clinical activity and safety of avelumab in patients with NEC G3 (WHO 2010), including "NET G3" who are progressive after first line chemotherapy.

DETAILED DESCRIPTION:
According to the WHO classification of 2010, Neuroendocrine neoplasms (NEN) are divided into well to moderately differentiated neuroendocrine tumors (NET), which are graded depending on their proliferation status into NET G1 (Ki67 index < 2%) and NET G2 (Ki67 2-20%), and into the poorly differentiated high grade neuroendocrine Carcinomas (NEC G3, ki67 > 20%), which - depending on their morphology - are subdivided into small cell as well as large cell NECs. The vast majority (60-90%) of patients with high grade NEC are metastasized at the time of diagnosis with distant metastases present in approximately two third of the patients.

G3 neuroendocrine neoplasia according to the WHO classification of 2010 are not a homogenous entity. Based on clinical and morphological criteria a differentiated subgroup with a Ki67 in the lower proliferative range (usually between 20-55%) which is unofficially termed "NET G3", can be subdivided from the more aggressive and undifferentiated "classical" NEC G3.

The prognosis of patients with metastatic NEC G3 is poor, and median overall survival has been reported to be 5 months with a 2-year survival rate of 11 % in the SEER data base for gastrointestinal NEC. In two large series of GEP-NEC, median survival was 12-19 months for patients with best available therapy (mainly platinum based chemotherapy) and as short as 1 month for those receiving only best supportive therapy. In contrast to the "classical" NEC G3 with a poorly differentiated morphology and a Ki 67 > 55%, NET G3 typically do not respond as well to a platinum based chemotherapy but a have a somewhat better prognosis with a 4-months longer median survival as compared to classical NEC G3. Therefore, according to current guidelines other treatment options like temozolomide based chemotherapy may be considered as a first line therapy in patients with differentiated "NET G3" .

There is a strong and unmet medical need for a novel and effective second line treatment option for these highly aggressive and rapidly progressing tumors. Considering the lack of any other established therapeutic option and the very limited efficacy of alternative second or third line chemotherapy in patients with NEC G3 (WHO 2010) who are progressive after a first-line chemotherapy, the availability of a novel therapeutic option with a significant clinical benefit (SD; PR; CR) in at least 30 % of the patients and with tolerable side effects would represent an important and clinical highly relevant break through in the treatment of these aggressive tumors.

There is a strong rationale for investigating PD-1/PD-L1 blockade in NEC G3 (WHO 2010). High grade NEC as well as LCNEC of the lung show a high mutational load, what is associated with a strong immunogenicity and a better response to an anti-PDL1/PD1 immunotherapy, and increased PDL1 expression has been demonstrated in high grade NEC. In intermediate NET the degree of T-cell tumor infiltration was associated with recurrence and survival and in a study with 80 patients with bronchopulmonary NEN including high grade NEC the expression of PD-L1 and PD-1 was associated with a worse prognosis. Evidence from phase 2 to 3 trials shows antiproliferative efficacy of an anti-PDL1/PD1 immunotherapy in high grade NECs. Furthermore, Merkel cell carcinomas, which are classified as high grade neuroendocrine tumors, are sucessfully treated with Avelumab.

Avelumab is a fully human antibody that binds PD-L1 and blocks the interaction between PD-L1 and PD-1. This removes the suppressive effect of PD-L1 on anti-tumor CD8+ T cells, resulting in restoration of cytotoxic T cell response.

Given the important role of PD-L1 in the suppression of T-cell responses, and the mode of action of avelumab which blocks the interaction between PD-L1 and its receptors, avelumab is being developed as a potential therapy for subjects with various tumors.

It is assumed that at least 20-30 % of patients with progressive disease after at least one first line chemotherapy will show a significant and clinically highly relevant benefit which is defined as an objective tumor response with complete remission (CR), partial remission (PR) or stable disease (SD) according to RECIST1.1.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥ 18 years
* Histologically proven neuroendocrine neoplasia NEC G3 (WHO 2010)
* One block or 20 slides (cut at 4 microns) of archival tumor tissue, if available, to perform biomarker assessment
* No curative option available
* Progressive disease within 9 months before study Initiation and after at least one chemotherapy (platinum based chemotherapy or STZ/TEM/DTIC based chemotherapy in NET G3)
* Presence of measurable disease as per RECIST1.1 criteria
* Physiologic function:

  * Hematologic: absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin ≥ 9 g/dL (may have been transfused)
  * Hepatic: total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range and AST and ALT levels ≤ 2.5 × ULN or AST and ALT levels ≤ 5 × ULN for subjects with documented metastatic disease to the liver)
  * Renal: estimated creatinine clearance ≥ 60 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
* Pregnancy and contraception:

  * Pregnancy test: Negative serum or urine pregnancy test at screening for women of childbearing potential.
  * Contraception: Highly effective contraception for both male and female subjects throughout the study and for at least 30 days for female and 90 days for male patients after avelumab treatment if the risk of conception exists.
* ECOG Performance Status 0 - 2
* Written informed consent: Signed and dated informed consent of the subject must be available before start of any specific trial procedures
* Ability of subject to understand nature, importance and individual consequences of clinical trial.

Exclusion Criteria:

* Merkel Cell carcinoma (MCC) or small cell lung cancer (SCLC)
* Typical or Atypical Carcinoid of the lung with a Ki67 < 20%
* Prior therapy with any antibody/drug targeting T-cell co-regulatory proteins (immune checkpoints)
* Neuroendocrine tumors that are potentially curable by surgery
* Major surgery within 4 weeks of initiation of study medication.
* TACE, TAE, SIRT or PRRT within 3 months of starting study treatment
* Patients pretreated with Interferon as last treatment line prior to study entry
* Concurrent anticancer treatment after the start of trial treatment (e.g., cyto-reductive therapy, TKI therapy, mTOR inhibitor therapy, radiotherapy [with the exception of palliative radiotherapy], immune therapy, or cytokine therapy except for erythropoietin or use of any investigational drug).
* Immunosuppressants: Current use of immunosuppressive medication, EXCEPT for the following:

  1. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
  2. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent;
  3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Prior organ transplantation, including allogeneic stem cell transplantation
* Active infection requiring systemic therapy
* HIV/AIDS: Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Hepatitis: Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
* Autoimmune disease: Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
* Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable
* Pregnancy or lactation
* Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Vaccination: Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines
* Hypersensitivity to study drug: Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3).
* Cardiovascular disease: Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Participation in other clinical trials during the present clinical trial or within the last 30 days or five terminal phase half-lives of the drug whichever is longer, prior to baseline (this also includes investigational formulation of market products).
* Medical or psychological conditions that would jeopardise an adequate and orderly completion of the trial.
* Patients, who are legally institutionalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
disease control rate (DCR) after 16 weeks of avelumab treatment | 16 weeks
  The primary endpoint is the disease control rate (DCR) after 16 weeks of avelumab treatment. DCR is defined as the percentage of subjects with a confirmed reduction in tumor size compared to baseline (complete response (CR) and partial response (PR)) as well as fulfilling the criteria for stable disease (SD) according RECIST1.1.

SECONDARY OUTCOMES:
disease control rate (DCR) on other assessments | 8, 24, 36, 48, 60 weeks
  Disease control rate (DCR) on other assessments. DCR is the proportion of patients with complete response, partial response and stable disease according to RECIST1.1.
Objective response rate (ORR) on every assessment | 8, 16, 24, 36, 48, 60 weeks
  Objective response rate (ORR) on every assessment. ORR is the proportion of patients with complete response (CR) or partial response (PR) according to RECIST1.1.
Best overall response (BOR) | 8, 16, 24, 36, 48, 60 weeks
  Best overall response (BOR). BOR is recorded from the start of the treatment until disease progression/recurrence according to RECIST1.1.
Duration of disease control | up to 1 year
  Duration of disease control: Duration of disease control is defined as the time from the first disease control (CR, PR, SD) to progression of disease (PD) according to RECIST1.1.
Time to response (TTR) | up to 1 year
  Time to response (TTR): TTR is the time from the first dose of trial medication to the first documentation of either complete response (CR) or partial response (PR) according to RECIST1.1.
Median Progression-free survival time (PFS) | up to 2 years
  Median Progression-free survival time (PFS). The time from first dose of trial medication to first documentation of objective tumor progression (PD) or to death due to any cause, whichever occurs first.
Overall survival (OS) and survival rate after 1 and 2 years | up to 2 years
  Overall survival (OS) and survival rate after 1 and 2 years: Overall survival is defined as the time from first dose of trial medication to date of death due to any cause. Survival rate is defined as rate of subjects surviving for at least 1 year or 2 years after first application of trial medication.
Quality of life (QoL) | 0, 8, 16, 24, 36, 48, 52, 60 weeks
  Quality of life (QoL) assessed by the EORTC QLQ-C30 questionnaire on Screening/Baseline, during Treatment on every assessment, on End of Treatment and on Safety FU visit
Incidence of adverse events (AEs) | 60 weeks
  Reporting of number and frequency of adverse Events (AEs) during treatment with avelumab and until Safety Follow

OTHER OUTCOMES:
assessment of serum levels in Chromatogranin A (CgA) | 0, 8, 16, 24, 36, 48, 60 weeks
  assessment of serum levels in Chromatogranin A (CgA) measured at time of tumor assessments
assessment of serum levels in Neuron specific enolase (NSE) | 0, 8, 16, 24, 36, 48, 60 weeks
  assessment of serum levels in and Neuron specific enolase (NSE) measured at time of tumor assessments
Tumor growth rate (TGR) | 0, 8, 16, 24, 36, 48, 60 weeks
  Tumor growth rate (TGR): TGR is the percentage change in tumor volume over one month
Tumor response according to irRECIST | 8, 16, 24, 36, 48, 60 weeks
  Tumor response according to irRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Matthias M Weber, MD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (4):
- Germany (4):
  - Poliklinik für Innere Medizin I Universitätsklinikum Halle, Halle
  - Nationales Centrum für Tumorerkrankungen Universitätsklinikum Heidelberg, Heidelberg
  - Schwerpunkt Endokrinologie und Stoffwechselerkrankungen Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Klinik für Innere Medizin, Abteilung Gastroenterologie Universitätsklinikum Gießen und Marburg, Marburg

IPD SHARING:
Plan to Share IPD: No